CLINICAL TRIAL: NCT01649986
Title: Additive Effects of Nutraceuticals to Non-pharmacologic Intervention to Improve Lipid Profile in the Real World Clinical Practice in European Countries - The PIN (Portugul Italy Nutraceutical) Study
Brief Title: Nutraceuticals to Improve Lipid Profile in European Countries
Acronym: PIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 450/2012/D
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; Non-pharmacologic prevention
MeSH Terms: conditions — Hyperlipidemias | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-pharmacologic intervention (Active Comparator): Patients assigned by their own general practitioner to have non-pharmacologic intervention and prevention strategies will be given details on lifestyle approaches and dietary strategies
  Interventions: Behavioral: Non-pharmacologic intervention
- Nutraceuticals (Active Comparator): Patients assigned by their own general practitioner to receive nutraceuticals, along with non-pharmacologic intervention and prevention strategies, will have for 1 year also 1 capsule/day containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg,
  Interventions: Drug: Nutraceuticals (Armolipid Plus)

INTERVENTIONS:
Behavioral: Non-pharmacologic intervention — Diet and physical exercise
  Other Names: Hypolipidemic non-pharmacologic intervention
  Arms: Non-pharmacologic intervention
Drug: Nutraceuticals (Armolipid Plus) — Patients assigned by their own general practitioner to receive nutraceuticals, along with non-pharmacologic intervention and prevention strategies, will have for 1 year also 1 capsule/day containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg,
  Other Names: Armolipid Plus, Rottapharm, Italy
  Arms: Nutraceuticals

SUMMARY:
Cardiovascular prevention include a class I indication to statins in addition to non-pharmacologic intervention and prevention strategies in patients deemed to be 'high risk' according to current scientific guidelines. In the real world, however, statin treatment is often discontinued due to side effects.

In addition, statins are not indicated in those subjects deemed to be 'low risk', in whom only non-pharmacologic intervention and prevention strategies are currently prescribed.

Along with non-pharmacologic intervention and prevention strategies, newer approaches to reduce cholesterol blood levels currently include nutraceuticals, which are compounds derived from foods with cholesterol lowering actions.

The primary objective of this study is twofold:

First, to prospectively compare in the real world clinical practice the efficacy and tolerability of non-pharmacologic intervention vs. the combination of non-pharmacologic intervention with a nutraceutical-based protocol in patients in whom statin treatment is not tolerated or is not indicated.

Second, to evaluate gender and race/ethnic differences in the hypolipidemic effects of a nutraceutical-based protocol among European countries.

DETAILED DESCRIPTION:
Cardiovascular prevention include a class I indication to statins in addition to non-pharmacologic intervention and prevention strategies in patients deemed to be 'high risk' according to current scientific guidelines. In the real world, however, statin treatment is often discontinued due to side effects.

In addition, statins are not indicated in those subjects deemed to be 'low risk', in whom only non-pharmacologic intervention and prevention strategies are currently prescribed.

Along with non-pharmacologic intervention and prevention strategies, newer approaches to reduce cholesterol blood levels currently include nutraceuticals, which are compounds derived from foods with cholesterol lowering actions.

In the real world clinical practice, however, it remains unclear if nutraceuticals yield additive therapeutic effects to non-pharmacologic intervention and prevention strategies in patients in whom statin treatment is not tolerated or is not indicated.

The primary objective of this study is twofold:

First, to prospectively compare in the real world clinical practice the efficacy and tolerability of non-pharmacologic intervention vs. the combination of non-pharmacologic intervention with a nutraceutical-based protocol in patients in whom statin treatment is not tolerated or is not indicated.

Second, to evaluate gender and race/ethnic differences in the hypolipidemic effects of a nutraceutical-based protocol among European countries.

Patients will be assigned at the discretion of their own general practitioner to receive for 1 year either non-pharmacologic intervention and prevention strategies or non-pharmacologic intervention and prevention strategies associated with a commercially available nutraceutical combined pill (1 capsule/day containing red yeast rice 200 mg, policosanol 10 mg, and berberine 500 mg).

ELIGIBILITY:
Inclusion Criteria:

* Class I indication to receive statin treatment but previous (<12 months) withdrawn of a statin due to side effects and unwilling to receive treatment with an alternative statin
* Class I indication to receive non-pharmacologic intervention and prevention strategies because of hyperlipidemia with 'low risk' classification
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment tolerability | Up to 12 months
  Reasons for treatment discontinuation

SECONDARY OUTCOMES:
Evaluation of drug effects on lipid and metabolic features | Up to 12 months
  Effects on lipid profile (total cholesterol, LDL cholesterol, triglycerides) and metabolic indexes (glucose levels, HOMA)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — Sapienza University
Locations (1):
- Sapienza University, Rome, Italy